CLINICAL TRIAL: NCT07392580
Title: A Single-Arm, Open-Label Study of Intralesional Treatment of Laryngeal Squamous Cell Carcinoma With Cisplatin
Brief Title: Intralesional Chemotherapy (IC): Cisplatin + Epinephrine
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, David Rosow, Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250847
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Laryngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Epinephrine; Endoscopy; Laryngectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cisplatin + Epinephrine Group (Experimental): Participants in this group will receive one (1) dose of intralesional chemotherapy (IC) treatment per week over a period of approximately 3 weeks. IC treatment will consist of combination cisplatin and epinephrine. Participants will then go to have endoscopic surgery for their disease.
  Total participation duration is approximately 16 months.
  Interventions: Drug: Cisplatin; Drug: Epinephrine injection; Procedure: Laryngeal Biopsy; Procedure: Endoscopic Surgery

INTERVENTIONS:
Drug: Cisplatin — Participants will be administered 1 mg/mL Cisplatin via intralesional injection in combination with Epinephrine injection therapy. Total treatment volume will determined by the volume of the tumor to be injected.
Drug: Epinephrine injection — Participants will be administered a 1:50,000 dilution of epinephrine via intralesional injection in combination with cisplatin therapy. The total treatment volume will determined by the volume of the tumor to be injected.
Procedure: Laryngeal Biopsy — At the time of the first intralesional chemotherapy (IC) dose, participants will have a biopsy of tumor tissue taken for standard of care (SOC) clinical activities. A portion of this sample will, if available, be banked for transcriptomic analysis.
Procedure: Endoscopic Surgery — Participants with early disease will go on to have endoscopic surgical resection of their cancer while participants with advanced disease will receive a total laryngectomy, after completion of intralesional chemotherapy (IC) therapy. Resected tissue collected at the time of the surgical procedure (either cordectomy or total laryngectomy) will also be banked for correlative studies.
  Other Names: Cordectomy; Laryngectomy

SUMMARY:
The purpose of this study is to determine the effects, good and bad, of injecting chemotherapy into recurrent laryngeal squamous cell carcinoma (SCC) tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 years and older.
2. Previously treated for laryngeal SCC with radiation.
3. Must have biopsy-proven recurrent cancer requiring surgical management. Note: if participants do not have an archived tissue sample available for review, they may undergo a biopsy procedure for collection of a fresh tissue sample for diagnostic confirmation and determination of further treatment. In this case, a fresh tumor sample would be used for diagnostic confirmation and trial eligibility. Please note, this biopsy would be considered a standard of care (SOC) procedure since it is being performed for disease management purposes regardless of participant enrollment in the trial.
4. Participants must be willing to undergo 3 weekly cycles of IC under local anesthesia prior to surgery.
5. Adequate hematologic, hepatic, and renal function tested within 6 weeks prior to the start of therapy (values must not be achieved with growth factors):

   1. Absolute neutrophil count (ANC) ≥ 1.0 × 10^9 cells /L.
   2. Hemoglobin ≥ 8.0 g/dL.
   3. Platelet count ≥ 50 × 10^9 platelets/L.
   4. Total bilirubin ≤ 1.5 × upper limit of normal (ULN).
   5. Alanine transaminase (ALT)/aspartate aminotransferase (AST) ≤ 3.0 ULN.
   6. Calculated creatinine clearance ≥ 45 mL/min by the Cockcroft-Gault Equation or the estimated glomerular filtration rate ≥ 45 mL/min/1.73 m2 using the Modification of Diet in Renal Disease formula.
6. Willingness to avoid pregnancy based on the criteria below:

   1. Woman of non-childbearing potential (ie, surgically sterile with a hysterectomy and/or bilateral oophorectomy OR ≥ 12 months of amenorrhea and at least 45 years of age).
   2. Woman of childbearing potential who has a negative urine or serum pregnancy test at screening and who agrees to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening and for at least 14 months after the last dose of trial intervention. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the participant and their understanding confirmed.

Exclusion Criteria:

1. Inability to tolerate awake, unsedated laryngeal procedures. Participants may opt to receive pre-procedure diazepam.
2. Participant unable to receive contrast.
3. Concurrent anticancer therapy (eg, chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, hormonal therapy, investigational therapy, or tumor embolization).
4. Receipt of anticancer medications or investigational drugs within the following intervals before the date of the first dose of trial intervention:

   1. < 10 weeks from completion of any radio- or toxin-immunoconjugates.
   2. < 4 weeks for immunotherapy.
   3. < 3 weeks for radiotherapy.
   4. < 2 weeks for any investigational agent or other anticancer medications.
   5. Steroids that are used for treatment of allergy or other underlying condition are permittable but not steroids started to treat cancer. Individuals receiving corticosteroids must be at a dose level ≤ 10 mg/day within 7 days of the trial intervention administration.
5. Inadequate recovery from toxicity and/or complications from a major surgery before starting therapy.
6. Current or previous other malignancy within 3 years of trial entry, except cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy.
7. Significant concurrent, uncontrolled medical condition, including, but not limited to, renal, hepatic, hematological, gastrointestinal (GI), endocrine, pulmonary, neurological, cerebral, or psychiatric disease.
8. Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment or exposure to a live vaccine within 30 days of dosing.
9. Known human immunodeficiency virus (HIV) infection or positivity on immunoassay. Note: HIV screening test is optional.
10. Current New York Heart Association Class II to IV congestive heart failure.
11. Uncontrolled or symptomatic arrhythmia or stroke in last 6 months, liver cirrhosis, or autoimmune disorder requiring immunosuppression or long-term corticosteroids (> 10 mg daily prednisone equivalent).
12. Currently pregnant or breastfeeding.
13. Any condition that would, in the Investigator's judgment, interfere with full participation in the trial, including administration of trial intervention and attending required trial visits; pose a significant risk to the patient; or interfere with interpretation of trial data.
14. Patients with impaired decision-making capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2031-04-01 (Estimated); Study Completion 2031-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall Pathologic Response Rate (OPRR) | About six (6) weeks
  Overall Pathologic Response Rate (OPRR) is defined as the number of participants with a complete response (CR) or partial response (PR) as the best response to intralesional chemotherapy (IC) treatment. ORRR will be assessed by pathology as percentage viable tumor on histopathology at time of surgical resection.

SECONDARY OUTCOMES:
Number of Participants Experiencing Treatment-Related Serious Adverse Events (SAEs) | About 18 weeks
  Incidence of treatment-related toxicity will be reported as the number of participants experiencing treatment-related serious adverse events (SAEs). SAEs will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0, per physician discretion.
Number of Participants Experiencing Treatment-Related Adverse Events (AEs) | About 18 weeks
  Incidence of treatment-related toxicity will be reported as the number of participants experiencing treatment-related adverse events (AEs). AEs will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0, per physician discretion.
Overall Radiographic Response Rate (ORRR) | About five (5) weeks
  Overall Radiographic Response Rate (ORRR) is defined as the number of participants with a complete responses (CR) or partial response (PR) as the best response to intralesional chemotherapy (IC) treatment by radiography (percent regression on computed tomography (CT) according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1, per physician discretion.
Overall Endoscopic Response Rate (OERR) | About five (5) weeks
  Overall Endoscopic Response Rate (OERR) is defined as the number of participants with a complete response (CR) or partial response (PR) as the best response to intralesional chemotherapy (IC) treatment by endoscopy (percent regression determined by blinded raters of pre- and post-IC endoscopy).

CONTACTS AND LOCATIONS:
Overall Officials: David Rosow, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No